CLINICAL TRIAL: NCT03592953
Title: Serious Games and Non Technical Skills Training: Are Scenarios Specifically Designed for Learning Non Technical Skills More Effective Than Baseline Scenario
Brief Title: Are Serious Games Scenarios Specifically Designed for Learning Non Technical Skills More Effective Than Baseline Scenarios in Soft Skills Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ilumens (Other)
Responsible Party: Principal Investigator, Daphne Michelet, Principal Investigator, Ilumens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Maccoy
Record Dates: First submitted 2018-07-05; First posted 2018-07-19 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Simulation Training
Keywords: Serious game; Post partum hemorrhage; Non technical skills
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Randomized trial with 3 groups: classical teaching, serious game with classical scenarios, serious game with specific scenarios
Who Masked: Outcomes Assessor
Masking Description: the primary endpoint is the scoring of non-technical skills on the video recording of the high fidelity simulation session. The raters are blinded of the allocation group of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Serious game Control group (Experimental): The participants spend on three different scenarios from the game PerinatSims; basic scenarios designed to train Technical Skills (management of post partum hemorrhage according to the algorithm).
  Interventions: Other: Serious game simulation training sessions
- Serious game Experimental group (Experimental): The participants spend on three "PerinatSims" scenarios in which "critical situations" have been implemented, aiming to mobilize some of the non-technical skills of the learners: situation awareness, decision making, communication...
  Interventions: Other: Serious game simulation training sessions
- Classical teaching group (No Intervention): the students received the classical teaching of postpartum hemorrhage management and a reminder of the algorithm before the high fidelity simulation session.

INTERVENTIONS:
Other: Serious game simulation training sessions — Each participant of the Serious game groups played 3 scenarios of "Perinatsims", a screen-based simulation on the management of a post partum hemorrhage. The serious game control group played basic scenarios and the experimental group played specific scenarios.
  Arms: Serious game Control group; Serious game Experimental group

SUMMARY:
The aim of the study is to assess if a training on post-partum hemorrhage management with serious game scenarios specifically designed to teach non technical skills improve non technical skills scoring in a high-fidelity simulation session.

DETAILED DESCRIPTION:
This study aims to answer the following problematic: How to improve the learning of Non Technical Skills (communication, teamwork, leadership ...) in simulation. This study tests non technical skills learning in a serious game on Postpartum Hemorrhage (PPH) management and the interest of specifically designed scenarios.

36 students in midwifery in 5th (and last) year will participate in the experiment. They will be randomized into 3 groups:

* Serious game Control group (12 participants): The participants spend on three different scenarios from the game "PerinatSims"; basic scenarios designed to train Technical Skills (management of post partum hemorrhage according to the algorithm).
* Serious game Experimental group (12 participants): The participants spend on three "PerinatSims" scenarios in which "critical situations" have been implemented, aiming to mobilize some of the non-technical skills of the learners: situation awareness, decision making, communication...
* Classical teaching group (12 participants): the students received the classical teaching of postpartum hemorrhage management and a reminder of the algorithm before the high-fidelity simulation session.

For the serious games groups, at the end of each scenario the participant has access to a debriefing of his technical skills, integrated into the game. At the end of the 3 scenarios, the participant has a debriefing with a simulation teacher.

Finally, each participant of the three groups will be asked to participate to a post partum hemorrhage scenario in High Fidelity simulation. This final award will enable us to validate the investigator's working hypothesis: to check if the non-technical skills mobilized during the sessions on the serious game PerinatSims have been acquired and are beneficial for the participants. A debriefing will be done at the end of the simulation.

The objective of this experiment is to assess if the type of scenario (with or without critical events) improves non-technical skills learning.

The evaluation tools will be the following:

* 3 hetero evaluation scales: Anesthetist's Non Technical Skills (ANTS), Observational Teamwork Assessment for Surgery (OTAS) and a checklist specially developped.
* Electrophysiology: Eye tracking (for the screen-based simulation), Heart rate monitor
* Auto evaluation scales: Flow scale, Stress scale (DASS), Leadership scale (BAT), Mental load scale (NASA TLX), Scale of technological acceptability (SUS)

The High Fidelity simulation will be evaluated according to the same tools outside the eye-tracking.

ELIGIBILITY:
Inclusion Criteria:

* Students in midwifery in 4th or 5th year (last year of the french curriculum)

Exclusion Criteria:

* Midwifery students who did not receive theoretical training on postpartum hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Non technical skills scoring with OTAS score | One year
  3 raters will evaluate participant on the video recording of the High fidelity simulation session with the help of the OTAS score (Observational Teamwork Assessment for Surgery). The total score is 30 points and is composed of 5 categories (/6 points each): communication, coordination, cooperation, leadership, situation awareness.

SECONDARY OUTCOMES:
Non technical skills scoring with a specific checklist for the assessment of non technical skills in post partum hemorrhage situation | One year
  3 raters will evaluate the participant on the video recording of the High fidelity simulation session with the help of a checklist specifically designed for the non-technical skills in the post partum hemorrhage. The total score is 24 and is divided in 6 categories (/4points each): communication, situation awareness, decision making,collaborative work, leadership, emotion management

CONTACTS AND LOCATIONS:
Locations (1):
- Ilumens, Paris Descartes University, Paris, France

IPD SHARING:
Plan to Share IPD: No